CLINICAL TRIAL: NCT06799676
Title: A Single-Arm, Multicenter, Open-Label Phase Ib/II Clinical Study on the Application of Linperlisib Plus the VRD Regimen in Newly Diagnosed Patients with Multiple Myeloma
Brief Title: A Phase Ib/II Clinical Study on the Application of Linperlisib Combined with the VRD Regimen in Newly Diagnosed Patients with Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuling Zhou (Other)
Responsible Party: Sponsor-Investigator, Fuling Zhou, PhD, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0101
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Newly Diagnosed Multiple Myeloma
Keywords: multiple myeloma; PI3Kδ inhibitor; Linperlisib
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- enrollment cohort (Experimental): Phase Ib ：Subjects will be administered Linperlisib orally at doses of 40 mg, 60 mg, or 80 mg once daily for 4 consecutive weeks, combined with the standard-dose VRD regimen. The dose-limiting toxicity (DLT) observation period is set at 28 days. If no DLT or other serious adverse events (SAEs) related to the investigational drug occur during the DLT observation period, the subject will proceed to subsequent treatment. In the absence of serious adverse events related to the investigational drug, the dose will be escalated to the next cohort based on the dose escalation principle.
  The Phase II expansion phase involves induction therapy with at least four cycles of Linperlisib at the recommended Phase II dose (RP2D) in combination with the VRD regimen. After completing four cycles of induction therapy, patients who meet the criteria for autologous hematopoietic stem cell transplantation (ASCT) will undergo the procedure. If a patient's therapeutic evaluation results in progressive disea
  Interventions: Drug: a combination treatment of Linperlisib and the VRD regimen

INTERVENTIONS:
Drug: a combination treatment of Linperlisib and the VRD regimen — Subjects will be administered Linperlisib orally at doses of 40 mg, 60 mg, or 80 mg once daily for 4 consecutive weeks, combined with the VRD regimen at standard doses. Subsequently, during the expansion phase, at least four cycles of Linperlisib at the recommended Phase II dose (RP2D) will be combined with the VRD regimen for induction therapy.

SUMMARY:
This study aims to evaluate the safety and efficacy of Linperlisib combined with the VRD regimen in the treatment of newly diagnosed patients with multiple myeloma. The study is divided into a Phase Ib dose exploration phase and a Phase II expansion phase.The Phase Ib dose exploration phase primarily aims to determine the recommended Phase II dose (RP2D) of Linperlisib based on dose-limiting toxicity (DLT). The Phase II expansion phase involves induction therapy using at least four cycles of Linperlisib at RP2D in combination with the VRD regimen. After completing four cycles of induction therapy, patients eligible for autologous hematopoietic stem cell transplantation (ASCT) will undergo the procedure. For patients whose therapeutic evaluation results in PD (progressive disease) or SD (stable disease), alternative treatment regimens will be considered based on their condition. After successful transplantation, 2-4 cycles of the original induction regimen will be used for consolidation therapy.The primary objective is to evaluate the proportion of patients achieving a very good partial response (VGPR) after four cycles of induction therapy with the Linperlisib combined VRD regimen.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients must be newly diagnosed with active multiple myeloma. 2. Patients must be between 18 and 65 years old and eligible for autologous hematopoietic stem cell transplantation (ASCT).

  3. Patients must have measurable disease, defined as follows:
* Any quantifiable serum monoclonal protein level (typically but not necessarily ≥0.5 g/dL of M-protein), and/or urinary light chain excretion >200 mg/24 hours.
* For oligosecretory or non-secretory multiple myeloma (MM), patients must have measurable plasmacytomas >2 cm confirmed by clinical examination or imaging (e.g., MRI, CT scan) or an abnormal free light chain (FLC) ratio (normal value: 0.26-1.65) with an involved FLC level ≥10 mg/dL.

  4. Patients must have an expected survival of ≥3 months. 5. Karnofsky Performance Status (KPS) score must be ≥60%. 6. Liver Function:
* Serum alanine aminotransferase (ALT) ≤3 times the upper limit of normal (ULN).
* Aspartate aminotransferase (AST) ≤3 times ULN.
* Direct bilirubin ≤2 mg/dL (34 µmol/L) within 14 days prior to randomization. 7. Neutrophil and Platelet Counts: Absolute neutrophil count (ANC) ≥1.0 × 10⁹/L within 14 days prior to randomization.Platelet count ≥75 × 10⁹/L (or ≥50 × 10⁹/L if >50% of bone marrow is involved with myeloma) within 14 days prior to randomization.

  8. Creatinine clearance (CrCl) ≥30 mL/min, measured or calculated using standard formulas (e.g., Cockcroft-Gault) within 7 days prior to randomization.

  9. Corrected serum calcium levels must be ≤14 mg/dL (3.5 mmol/L). 10. Left ventricular ejection fraction (LVEF) must be ≥40%. Two-dimensional transthoracic echocardiography (ECHO) is the preferred method for assessment. If ECHO is unavailable, a multigated acquisition scan (MUGA) is acceptable.

  11. Patients must be able to understand and voluntarily sign the informed consent form.

  12. Women with childbearing potential must agree to undergo pregnancy testing and use contraception.

  13. Male subjects must agree to use contraception.

Exclusion Criteria:

* 1. Patients who have previously received anti-myeloma therapy, except for radiotherapy, bisphosphonates, or a single short course of steroids (≤40 mg/day of dexamethasone equivalent for up to 4 days).

  2. Non-secretory MM patients, unless they have abnormal serum free light chains or a measurable plasmacytoma with a minimum maximum diameter >2 cm.

  3. Patients who do not meet the eligibility criteria for autologous stem cell transplantation.

  4. Women who are pregnant or breastfeeding. 5. Acute active infections requiring treatment (ongoing use of systemic antibiotics, antiviral, or antifungal agents) within 14 days prior to randomization.

  6. Patients with known human immunodeficiency virus (HIV) infection. 7. Active hepatitis A, B, or C infection. 8. Patients with the following cardiac conditions within 4 months prior to randomization:
* Unstable angina or myocardial infarction.
* New York Heart Association (NYHA) Class III or IV heart failure.
* Uncontrolled angina.
* Severe coronary artery disease.
* Severe ventricular arrhythmias.
* Sick sinus syndrome.
* Acute ischemia.
* Electrocardiographic evidence of Grade 3 conduction abnormalities, unless the patient has a pacemaker.

  9. Severe neuropathy (Grade 3-4 or Grade 2 with pain) as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC) Version 4.0 within 14 days prior to randomization.

  10. Known allergy to any of the investigational drugs. 11. Patients with contraindications to required concomitant medications or supportive therapies, including hypersensitivity to all anticoagulants, antiplatelets, or antiviral agents, or intolerance to hydration due to pre-existing pulmonary or cardiac impairment.

  12. Any other clinically significant disease or condition that, in the investigator's opinion, could interfere with protocol adherence or the patient's ability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | At the end of Cycle 4 (each cycle is 28 days)
  The primary objective is to determine the recommended Phase II dose (RP2D) of Linperlisib based on dose-limiting toxicity (DLT).
VGPR Rate | At the end of Cycle 4 (each cycle is 28 days)
  The very good partial response (VGPR) rate is evaluated based on the 2016 International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Complete remission rate | At the end of Cycle 4 (each cycle is 28 days)
  Bone marrow primitive cells <5%, no primitive cells with Auer vesicles, no primitive cells in the peripheral blood, no extramedullary leukaemia, neutrophil count ≥1.0×109/L, platelet count ≥100×109/L
Overall survival | Time from the patient's first dose of medication to death from any cause (Assessment of up to 100 months from the date of randomisation to the date of first recorded progress or the date of death from any cause, whichever comes first)
  The time from the patient's first dose of medication to the time of death from any cause.
Progression-Free Survival (PFS) | Time from the patient's first dose of medication to death from any cause (Assessment of up to 100 months from the date of randomisation to the date of first recorded progress or the date of death from any cause, whichever comes first)
  The length of time during and after treatment that a patient lives without any signs of disease progression, assessed after completing induction therapy, ASCT, and consolidation therapy.
Incidence of adverse events | At the end of Cycle 4 (each cycle is 28 days)
  Incidence of adverse events, e.g., GI adverse reactions, cardiotoxicity, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fuling Zhou, Study Director — Zhongnan Hospital
Locations (3):
- China (3):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xianning Central Hospital, Xianning, Hubei

IPD SHARING:
Plan to Share IPD: No